CLINICAL TRIAL: NCT00995475
Title: A Proof of Concept Study to Evaluate the Dose Response for the Systemic Benefit Risk Ratio of Inhaled Fluticasone Propionate in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MEN001
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2019-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled corticosteroid, Then placebo (Experimental): FP 250μg per actuation pMDI one puff twice daily (total daily dose 500μg) for two weeks then FP 250μg per actuation pMDI four puffs twice daily (total daily dose 2000μg) for two weeks. After a washout period of 2 weeks, they then received FP matched placebo pMDI one puff twice daily for two weeks then FP four puffs twice daily for two weeks.
  Interventions: Drug: Fluticasone propionate; Drug: Placebo
- Placebo control, Then inhaled corticosteroid (Placebo Comparator): FP matched placebo pMDI one puff twice daily for two weeks then FP four puffs twice daily for two weeks. After a washout period of 2 weeks, they then received FP 250μg per actuation pMDI one puff twice daily (total daily dose 500μg) for two weeks then FP 250μg per actuation pMDI four puffs twice daily (total daily dose 2000μg) for two weeks.
  Interventions: Drug: Fluticasone propionate; Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate
Drug: Placebo

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major worldwide problem.Steroids inhalers are now an established treatment for COPD. Inhaled steroids can have a number of bad effects including suppression of the adrenal glands because of absorption. A previous study in patients with COPD.

C-reactive Protein (CRP) is a peptide produced in the liver in response to inflammation. Elevated circulating levels of CRP are associated with heart conditions. High levels of CRP have also been found in patients with COPD. In some studies, steroid inhalers have reduced CRP levels, and that of other inflammatory mediators, in patients with COPD. It is unknown whether this reflects a reduction in lung inflammation or an effect of systemically absorbed corticosteroid.

It is proposed to investigate the link between inhaled corticosteroid and serum CRP, lung inflammation (measured by exhaled nitric oxide) and systemic absorption of steroids.

ELIGIBILITY:
Inclusion Criteria:

* Current or ex-smokers
* Aged over 50years
* FEV1/FVC ratio <0.7
* FEV1<80% predicted
* Improvement in FEV1 following short acting beta-agonist not greater than 15% and 200ml.

Exclusion Criteria:

* Diagnosis of asthma, bronchiectasis or ABPA
* Inability to perform study procedures or give informed consent
* Known sensitivity to trial medications

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

REFERENCES:
- [Result] Williamson PA, Menzies D, Clearie KL, Vaidyanathan S, Lipworth BJ. Dose-response for inhaled fluticasone on airway and systemic inflammation in COPD. Eur Respir J. 2011 Jan;37(1):206-9. doi: 10.1183/09031936.00062210. No abstract available. PMID 21205715

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomised, double blind placebo controlled cross over trial design will be used. Following a two-week steroid tapering process and a two-week run in period, two randomised treatment periods will follow. Each will be one month in duration and will be separated by a two-week wash-out period.
Groups:
- Inhaled Corticosteroid One Month: FP 250μg per actuation pMDI one puff twice daily (total daily dose 500μg) for two weeks then FP 250μg per actuation pMDI four puffs twice daily (total daily dose 2000μg) for two weeks. Then two-week washout before placebo.
  Fluticasone propionate
- Placebo Control One Month: FP matched placebo pMDI one puff twice daily for two weeks then FP four puffs twice daily for two weeks. Then two-week washout before FP.
  Placebo
Period: First Intervention
Arm/Group | Inhaled Corticosteroid One Month | Placebo Control One Month
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Wash-out Two Week
Arm/Group | Inhaled Corticosteroid One Month | Placebo Control One Month
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Inhaled Corticosteroid One Month | Placebo Control One Month
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a cross over trial in which 18 participants completed the trials.
Groups:
- Inhaled Corticosteroid, Then Placebo or Vice Versa: FP 250μg per actuation pMDI one puff twice daily (total daily dose 500μg) for two weeks then FP 250μg per actuation pMDI four puffs twice daily (total daily dose 2000μg) for two weeks.
  Then 2 weeks of wash-out.
  Then followed by FP matched placebo pMDI one puff twice daily for two weeks then FP four puffs twice daily for two weeks.
Arm/Group | Inhaled Corticosteroid, Then Placebo or Vice Versa
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: CRP
Description: C-reactive protein
Time Frame: 4 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Groups:
- Inhaled Corticosteroid: FP 250μg per actuation pMDI one puff twice daily (total daily dose 500μg) for two weeks then FP 250μg per actuation pMDI four puffs twice daily (total daily dose 2000μg) for two weeks.
  Fluticasone propionate
- Placebo Control: FP matched placebo pMDI one puff twice daily for two weeks then FP four puffs twice daily for two weeks.
  Placebo
Arm/Group | Inhaled Corticosteroid | Placebo Control
Number analyzed (Participants) | 18 | 18
mg/L | 2.9 [1.3 to 6.4] | 2.0 [1.1 to 3.4]

2. Secondary Outcome: Alveolar Nitric Oxide
Time Frame: 4 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: ppb
Arm/Group | Inhaled Corticosteroid | Placebo Control
Number analyzed (Participants) | 18 | 18
ppb | 1.7 [1.2 to 2.4] | 3.1 [2.6 to 3.8]

3. Secondary Outcome: OUCC
Description: Overnight urinary cortisol creatinine ratio
Time Frame: 4 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/mmol
Arm/Group | Inhaled Corticosteroid | Placebo Control
Number analyzed (Participants) | 18 | 18
nmol/mmol | 2.7 [1.6 to 4.6] | 8.8 [6.7 to 11.4]

ADVERSE EVENTS:
Arm/Group | Inhaled Corticosteroid | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes